CLINICAL TRIAL: NCT00968825
Title: A Phase 2, Double-Blind, Randomized, Parallel-Group, Controlled, Multi-Center Study to Evaluate the Efficacy and Safety of a Single Administration of RT001, a Botulinum Toxin Type A Topical Gel, for the Treatment of Moderate to Severe Lateral Canthal Lines in Adults
Brief Title: Safety and Efficacy Study of RT001 to Treat Moderate to Severe Lateral Canthal Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RT001-CL012LCL
Record Dates: First submitted 2009-08-27; First posted 2009-08-31 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-10

CONDITIONS: Lateral Canthal Lines; Crow's Feet; Facial Wrinkles
Keywords: Lateral Canthal Lines; Crow's Feet; Facial Wrinkles
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose D (Active Comparator): RT001
  Interventions: Drug: Botulinum Toxin Type A
- Dose E (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum Toxin Type A — RT001 (Botulinum Toxin Type A Topical Gel) Dose D applied topically at Baseline (Day 0) to the lateral canthal lines
  Arms: Dose D
Drug: Placebo — Placebo (Dose E) applied topically at Baseline (Day 0) to the lateral canthal lines
  Arms: Dose E

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a single administration of RT001 compared to placebo gel for the treatment of moderate to severe lateral canthal lines.

DETAILED DESCRIPTION:
This is a double-blind, randomized, parallel-group, controlled, multi-center study to evaluate the efficacy and safety of a single administration of RT001 compared to placebo applied as a bilateral application in at least 72 subjects with moderate to severe Lateral Canthal Lines. Subjects will be randomized within each site to 1 of 2 treatment groups in a 1:1 ratio. The efficacy and safety of RT001 compared to placebo will be evaluated. Study follow-up visits will occur at Weeks 2, 4 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, 30 to 60 years of age
* Bilateral lateral canthal lines rated as moderate or severe based on the Investigator Global Assessment - Lateral Canthal Lines Rest and Investigator Global Assessment - Lateral Canthal Lines Smile Severity Scales
* Willing to refrain from receiving facial fillers, laser treatments, use of any product that affects skin remodeling or a product that may cause an active dermal response in the treatment area beginning at Screening and through End of Study (Week 6)
* Women of childbearing potential must be practicing and willing to continue to use an effective method of birth control during the course of the study

Exclusion Criteria:

* Any neurological condition that may place the subject at increased risk with exposure to Botulinum Toxin Type A, including peripheral motor neuropathic diseases such as amyotrophic lateral sclerosis and motor neuropathy, and euromuscular junctional disorders
* Muscle weakness or paralysis in the area receiving study treatment
* Active skin disease or irritation at the treatment areas
* Eyelid ptosis, excessive dermatochalasis, deep dermal scarring or inability to substantially lessen the lateral canthal lines to be treated by physically spreading them apart
* Use of prescription retinoid products during the past 3 months prior to Screening
* Chemical peel (medium depth or deeper) during the past 9 months prior to Screening
* Undergone any procedures that may affect the lateral canthal region such as: periorbital surgery, brow left or related procedures, laser skin resurfacing or soft tissue augmentation (upper half of face) during the past 12 months prior to Screening
* Screening electrocardiogram (ECG) that is abnormal or clinically significant or any history of hypokalemia, torsade de pointe, unstable angina, myocardial infarction or congestive heart failure or family history of prolonged QT
* Previous treatment with Botulinum Toxin Type A in the face area
* Previous treatment with greater than 200 U Botulinum Toxin Type A anywhere else in the body within the last 6 months prior to Screening
* Concurrent use of aminoglycoside antibiotics, or other agents that might interfere with neuromuscular transmission starting at Screening
* Use of a topical steroid on either of the treatment areas or use of medications that suppress the immune system 30 days prior to Screening and continuing through End of Study (Week 6)
* Clinically significant laboratory values at Screening

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The number of subjects classified as exhibiting improvement via the Investigator Global Assessment of Lateral Canthal Line Severity at Rest from Baseline (Day 0) to Week 4; incidence of treatment emergent AEs | Week 4

SECONDARY OUTCOMES:
The number of subjects classified as exhibiting improvement via the Investigator Global Assessment of Lateral Canthal Line Severity at Rest and Smile from Baseline (Day 0) to Week 4 and Baseline (Day 0) to Week 6; incidence of treatment emergent AEs | Week 4 and Week 6

CONTACTS AND LOCATIONS:
Locations (1):
- RGG, Inc, San Francisco, California, United States